CLINICAL TRIAL: NCT04459208
Title: Randomized Comparison of Catheter-based Strategies for Interventional Access Site Closure During Transfemoral Transcatheter Aortic Valve Implantation
Acronym: CHOICE-CLOSURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helios Health Institute GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0191
Record Dates: First submitted 2020-06-26; First posted 2020-07-07 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Aortic Valve Stenosis
Keywords: Vascular access site closure; Transcatheter aortic valve implantation; Vascular closure device; Vascular access-site injury
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Investigator-initiated, single-center, prospective, open-label randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manta (Active Comparator): plug-based vascular closure
  Interventions: Device: Manta
- ProGlide (Active Comparator): suture-based vascular closure
  Interventions: Device: ProGlide

INTERVENTIONS:
Device: Manta — plug-based vascular closure
  Arms: Manta
Device: ProGlide — suture-based vascular closure
  Arms: ProGlide

SUMMARY:
The aim of the study is to evaluate the clinical efficacy of 2 different vascular closure device (VCD) strategies during transfemoral transcatheter aortic valve implantation (TAVI). The study hypothesizes that the choice of one over the other VCD in patients undergoing transfemoral TAVI may demonstrate relevant differences in the rate of peri-procedural complications and effectiveness of vascular closure.

DETAILED DESCRIPTION:
Use of a plug-based VCD in patients undergoing transfemoral TAVI as compared to a suture-based VCD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an indication for transfemoral TAVI as judged by the local heart team.
2. Transfemoral access route and a commercially-available transcatheter aortic valve is selected by the local heart team.
3. The patient is willing to provide written informed consent and comply with protocol- specified follow-up evaluations.

Exclusion Criteria:

1. Vascular access site anatomy not suitable for percutaneous vascular closure.
2. Vascular access site complications prior to the TAVI procedure.
3. Known allergy or hypersensitivity to any VCD component.
4. Unstable active bleeding/ bleeding diathesis or significant unmanageable anemia.
5. Absence of computed tomographic data of the access site before the procedure.
6. Systemic infection or a local infection at or near the access site.
7. Life expectancy of less than 6 months due to non-cardiac conditions.
8. Patient cannot adhere to or complete the investigational protocol for any reason.
9. Pregnant or nursing subjects.
10. Participation in any other interventional trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-08-04 (Actual)

PRIMARY OUTCOMES:
Rate of in-hospital access-site or access-related vascular injury according to the VARC-2 definition | up to 7 days
  Rate of in-hospital access-site or access-related vascular injury according to the VARC-2 definition

SECONDARY OUTCOMES:
Rate of access-site or access-related vascular injury | 30 days
  Rate of access-site or access-related vascular injury
Rate of major access-site or access-related vascular injury | up to 7 days and at 30 days
  Rate of major access-site or access-related vascular injury
Rate of minor access site or access-related vascular injury | up to 7 days and at 30 days
  Rate of minor access site or access-related vascular injury
Rate of access-site or access-related vascular injury, access-site or access-related bleeding and VCD failure according to VARC-2 criteria | up to 7 days and at 30 days)
  Rate of access-site or access-related vascular injury, access-site or access-related bleeding and VCD failure according to VARC-2 criteria
all-cause death | up to 7 days and 30-day
  all-cause death
death attributed to access-site or access-related complications | up to 7 days and 30-day
  death attributed to access-site or access-related complications
Unplanned vascular surgery and / or use of endovascular stent or stent-graft or other endovascular interventions at the puncture site | up to 7 days
  Unplanned vascular surgery and / or use of endovascular stent or stent-graft or other
access-site or access-related disabling/life- threatening bleeding according to BARC | up to 7 days and 30-day
  access-site or access-related disabling/life- threatening bleeding according to BARC
access-site or access-related major bleeding according to BARC | up to 7 days and 30-day
  access-site or access-related major bleeding according to BARC
access-site or access-related minor bleeding according to BARC | up to 7 days and 30-day
  access-site or access-related minor bleeding according to BARC
Need for blood transfusion for access-site or access-related bleeding or vascular complications | up to 7 days
  Need for blood transfusion for access-site or access-related bleeding or vascular complications
Total number of blood transfusions because of access-site or access-related bleeding | up to 7 days
  Total number of blood transfusions because of access-site or access-related bleeding
Rate of vascular closure device success, defined as the ability of a closure device strategy to obtain hemostasis | 24 hours
  Rate of vascular closure device success, defined as the ability of a closure device strategy to obtain hemostasis
Rate of vascular closure device failure, defined as failure of a closure device strategy to achieve hemostasis with the need for an alternative treatment | 24 hours
  Rate of vascular closure device failure, defined as failure of a closure device strategy to achieve hemostasis with the need for an alternative treatment
Length of postprocedural hospital stay | up to 7 days
  Length of postprocedural hospital stay
Time to hemostasis, defined as the time from VCD application to complete hemostasis | 24 hours
  Time to hemostasis, defined as the time from VCD application to complete hemostasis
Need and number of additional unplanned VCDs | 24 hours
  Need and number of additional unplanned VCDs
Percent diameter stenosis of vascular access vessel on post-procedural angiography | 24 hours
  Percent diameter stenosis of vascular access vessel on post-procedural angiography

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdel-Wahab, PD Dr., Principal Investigator — Herzzentrum Leipzig GmbH
Locations (1):
- Herzzentrum Leipzig, Leipzig, Germany

REFERENCES:
- [Derived] Abdel-Wahab M, Hartung P, Dumpies O, Obradovic D, Wilde J, Majunke N, Boekstegers P, Muller R, Seyfarth M, Vorpahl M, Kiefer P, Noack T, Leontyev S, Sandri M, Rotta Detto Loria J, Kitamura M, Borger MA, Funkat AK, Hohenstein S, Desch S, Holzhey D, Thiele H; CHOICE-CLOSURE Investigators. Comparison of a Pure Plug-Based Versus a Primary Suture-Based Vascular Closure Device Strategy for Transfemoral Transcatheter Aortic Valve Replacement: The CHOICE-CLOSURE Randomized Clinical Trial. Circulation. 2022 Jan 18;145(3):170-183. doi: 10.1161/CIRCULATIONAHA.121.057856. Epub 2021 Nov 5. PMID 34738828